CLINICAL TRIAL: NCT06162273
Title: Comparing the Efficacy and Safety of IBD Stent of Shenzhen Xianjian Company and IBE Stent of American Gore Company for Reconstruction of Internal Iliac Artery in Abdominal Aortic Aneurysm/Iliac Aneurysm Repair
Brief Title: An Exploratory Study of Iliac Artery Branch Stent for Internal Iliac Artery Reconstruction in Abdominal Aortic Aneurysm/Iliac Aneurysm Repair
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: The SIRI study
Record Dates: First submitted 2023-12-01; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Aortic Aneurysm, Abdominal; Iliac Aneurysm
Keywords: Iliac artery branch stent; Patency rate; Internal iliac artery
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Iliac Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD stent of Shenzhen Xianjian Company and IBE stent of American Gore company: Patients underwent endovascular treatment for reconstruction of internal iliac artery in abdominal aortic aneurysm/iliac aneurysm repair. The lesion will be treated by IBD stent of Shenzhen Xianjian Company and IBE stent of American Gore Company.
  Interventions: Device: IBD stent of Shenzhen Xianjian Company and IBE stent of American Gore company

INTERVENTIONS:
Device: IBD stent of Shenzhen Xianjian Company and IBE stent of American Gore company — Patients underwent endovascular treatment for reconstruction of internal iliac artery in abdominal aortic aneurysm/iliac aneurysm repair. The lesion will be treated by IBD stent of Shenzhen Xianjian Company and IBE stent of American Gore Company.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of IBD stent of Shenzhen Xianjian Company and IBE stent of American Gore company in the treatment of abdominal aortic aneurysm/iliac aneurysm reconstruction of internal iliac artery

DETAILED DESCRIPTION:
This study is a prospective observational exploratory cohort study without a control group. As a single-group target value validation study, the main evaluation indicator is the primary patency rate one year after surgery. As an exploratory study, considering the enrollment ability to facilitate data analysis, 40 subjects are enrolled in the final study, and 20 are expected to be included in each study. All enrolled patients will be followed for 12 months for CTA to assess primary patency. Telephone follow-up was conducted at 1, 3, 6, and 12 months for adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with iliac aneurysms combined with or without abdominal aortic aneurysms and internal iliac arteries reconstructed with iliac branch stents;
2. Male or female ≥18 years old, ≤85 years old;
3. Life expectancy > 2 years;
4. The patient signed the informed consent voluntarily and was able to comply with the treatment plan and complete the follow-up and examination as planned.

Exclusion Criteria:

1. Fungal or ruptured aneurysm
2. Known complications of thoracic aortic aneurysm require interventional treatment
3. American Association of Anesthesiologists (ASA) Grade V
4. Creatinine > 2.5mg/dL or dialysis patients
5. NYHA Grade IV heart failure
6. Intercalation, severe calcification, or anchoring area with thrombosis
7. Severe curvature or narrowing of the iliac and/or femoral arteries, resulting in difficulty in stent delivery
8. Conduct another device or drug study within 1 year of treatment
9. Systemic infection
10. Combined with connective tissue disease
11. Known history of drug use
12. Known allergies or allergies to equipment materials

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with iliac aneurysms/abdominal aortic aneurysms requiring iliac branch stents
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12-month
  CTA showed patency of the preserved internal iliac artery.

SECONDARY OUTCOMES:
New hip lameness | 12-month
  New hip lameness is defined as new hip claudication in the lateral body treated with an iliac artery branch stent.
Internal leakage | 12-month
  Internal leakage is defined as any type of internal leakage that occurs during the follow-up period.
Aneurysmal enlargement | 12-month
  Aneurysm enlargement is defined as having a larger aneurysm diameter during follow-up than before surgery.
Aneurysm rupture | 12-month
  Ruptured aneurysms is defined as ruptured abdominal aortic aneurysms or iliac aneurysms that occurrs during follow-up.
Secondary patency | 12-month
  Secondary patency is defined as maintaining patency in the target vessel after a repeat intervention to correct complete occlusion in the treated arterial segment.
Secondary endovascular repair surgery | 12-month
  Secondary endovascular repair is defined as secondary surgical intervention that occurrs during follow-up due to adverse events such as internal leakage and distal limb ischemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China